CLINICAL TRIAL: NCT03059797
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Clinical Trial to Compare the Efficacy and Safety of Anlotinib Versus Placebo in Patients With Small Cell Lung Cancer(ALTER1202)
Brief Title: Study of Anlotinib in Patients With Small Cell Lung Cancer (ALTER1202)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALTN-12-II
Record Dates: First submitted 2017-02-16; First posted 2017-02-23 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — anlotinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anlotinib (Experimental): Anlotinib Day 1 to day 14 followed by 7 days off treatment in a 21-day cycle
  Interventions: Drug: Anlotinib
- Placebo (Placebo Comparator): Placebo Day 1 to day 14 followed by 7 days off treatment in a 21-day cycle
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anlotinib — Anlotinib Day 1 to day 14 followed by 7 days off treatment in a 21-day cycle
  Arms: Anlotinib
Drug: Placebo — Placebo Day 1 to day 14 followed by 7 days off treatment in a 21-day cycle
  Arms: Placebo

SUMMARY:
To compare the effects and safety of Anlotinib with placebo in patients with small cell lung cancer(SCLC).

ELIGIBILITY:
Inclusion Criteria:

* Histological documentation of small cell lung cancer
* Advanced small cell lung cancer who had at least two chemotherapy regimens,at least one measurable lesion (by RECIST1.1)
* 18-75 years,ECOG PS:0-2,Life expectancy of more than 3 months
* Main organs function is normal
* Women of childbearing potential should agree to use and utilize an adequate method of contraception (such as intrauterine device，contraceptive and condom) throughout treatment and for at least 6 months after study is stopped；the result of serum or urine pregnancy test should be negative within 7 days prior to study enrollment，and the patients required to be non-lactating；Man participants should agree to use and utilize an adequate method of contraception throughout treatment and for at least 6 months after study is stopped
* Patients should participate in the study voluntarily and sign informed consent

Exclusion Criteria:

* Patients who have been used anlotinib
* Patients who have been used targeted drugs(such as sunitinib,bevacizumab,endostar),Immune targeted drugs
* 4 weeks or less from the last cytotoxic therapy, radiation therapy or surgery
* Patients whose primary lesion with active bleeding within 4 months
* Carcinomatous meningitis
* Patients who known to the central nervous system
* Patients with factors that could affect oral medication (such as dysphagia，chronic diarrhea, intestinal obstruction etc.)
* Patients with any severe and/or unable to control diseases，including：

  1. Blood pressure unable to be controlled ideally(systolic pressure≥150 mmHg，diastolic pressure≥100 mmHg);
  2. Patients with Grade 1 or higher myocardial ischemia, myocardial infarction or malignant arrhythmias(including QTc≥450ms(male),QTc≥470ms（female）) and patients with Grade 1 or higher congestive heart failure (NYHA Classification);
  3. Patients with active or unable to control serious infections;
  4. Patients with cirrhosis, decompensated liver disease, or active hepatitis;
  5. Patients with poorly controlled diabetes (fasting blood glucose(FBG)>10mmol/L)
  6. Urine protein ≥ ++，and 24-hour urinary protein excretion>1.0 g confirmed;
* Patients with non-healing wounds or fractures
* Patients with arterial or venous thromboembolic events occurred within 6 months, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism
* Patients with drug abuse history and unable to get rid of or Patients with mental disorders
* Imaging showed tumors have involved important blood vessels or by investigators determine likely during the follow-up study and cause fatal hemorrhage
* History of immunodeficiency
* Patients with concomitant diseases which could seriously endanger their own safety or could affect completion of the study according to investigators' judgment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-05-06 (Actual)

PRIMARY OUTCOMES:
Progress free survival (PFS) | From randomization，each 42 days up to PD or death(up to 24 months)

SECONDARY OUTCOMES:
Overall Survival (OS) | From randomization until death (up to 24 months)
Objective Response Rate (ORR) | each 42 days up to intolerance the toxicity or PD (up to 24 months)
Disease Control Rate (DCR) | each 42 days up to intolerance the toxicity or PD (up to 24 months)
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Until 30 day safety follow-up visit (up to 24 months)

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The 307th Hospital of Chinese People's Liberation Army, Beijing, Beijing Municipality
  - Guangdong General Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Harbin medical university affiliated tumor hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jilin Cancer Hospital, Changchun, Jilin
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Linyi Cancer Hospital, Linyi, Shandong
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gong J, Wan Q, Shang J, Qian X, Su D, Sun Z, Liu G. Cost-Effectiveness Analysis of Anlotinib as Third- or Further-Line Treatment for Relapsed Small Cell Lung Cancer (SCLC) in China. Adv Ther. 2021 Oct;38(10):5116-5126. doi: 10.1007/s12325-021-01889-2. Epub 2021 Aug 21. PMID 34417989
- [Derived] Zhang C, Wang J, Wang X, Meng Z, Cheng Y, Li K. Peripheral blood indices to predict PFS/OS with anlotinib as a subsequent treatment in advanced small-cell lung cancer. Cancer Biol Med. 2021 Jul 24;19(8):1249-58. doi: 10.20892/j.issn.2095-3941.2020.0727. PMID 34302324
- [Derived] Cheng Y, Wang Q, Li K, Shi J, Liu Y, Wu L, Han B, Chen G, He J, Wang J, Lou D, Yu H, Wang S, Qin H, Li X. Anlotinib vs placebo as third- or further-line treatment for patients with small cell lung cancer: a randomised, double-blind, placebo-controlled Phase 2 study. Br J Cancer. 2021 Aug;125(3):366-371. doi: 10.1038/s41416-021-01356-3. Epub 2021 May 18. PMID 34006926